CLINICAL TRIAL: NCT05011071
Title: The Alberta BLOOM Premature Child Study: Impact of the Microbiome on the Clinical Course and Health Outcomes of Premature Children
Brief Title: The Alberta BLOOM Premature Child Study
Acronym: BLOOM-PCS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Marie-Claire Arrieta, Assistant Professor, University of Calgary
Other Study IDs: REB20-1442
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Infant Conditions; Infant, Premature, Diseases; Asthma; Asthma in Children; Infant ALL; Allergy
Keywords: Microbiota; Microbiome; Gastrointestinal Microbiome; immunobiome
MeSH Terms: conditions — Infant, Premature, Diseases; Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Infant Samples: fecal, urine, hair, blood, nasopharyngeal swab. Maternal Samples: fecal and expressed breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, observational clinical cohort study involving 405 children born premature (at less than 37 weeks gestation) and their mother/parent/guardian. The purpose of the study is to investigate how the microbiome (the collection of microbes in a biological site) of children develops over the first years of life and its associations with the risk of childhood health outcomes including allergies and asthma. The study will also examine how perinatal factors associate with patterns of microbiome development, and their effects on the microbiome, metabolome (the collection of metabolites in a biological sample) and immune development of this population in the first years of life.

DETAILED DESCRIPTION:
Premature birth (birth before 37 weeks of pregnancy) occurs in about 1 in 10 pregnancies. When infants are born prematurely their gut is not as developed. One important factor in gut health is the large community of microbes (tiny living things such as bacteria) that live on the human body called the microbiome. Recent studies have shown that premature infants are more likely to experience changes to their gut microbiome that are associated with health issues, such as asthma and allergies. However, the specific microbiome features of children born preterm and the role of their microbiome in disease risk and childhood health is not well understood. The Alberta BLOOM Premature Child Study (PCS) investigates how the microbiome and immune health of premature children develops over the first years of life and its associations with the risk of childhood health outcomes. BLOOM-PCS will also study how the microbiome of children born premature differs from the microbiome in the term population.

The type of microbes that are present in the infant's gut in the first months of life have a major impact on the microbiome that will form during childhood. There are many environmental factors during pregnancy, birth and the first months of life that can impact an infant's microbiome development. Factors such as diet, exposure to antibiotics, surgical procedures, and mode of delivery can strongly affect early microbiome development. This study will investigate how these factors influence the types of early microbes present in preterm infants.

This study hypothesizes that specific microbial patterns, trajectories and/or metabolites will be significantly associated with single or a combination of perinatal maternal and/on infant factors. Also, that microbial alterations resulting from preterm birth contributes to the allergy and asthma outcomes in infants through immune mechanisms.

ELIGIBILITY:
Inclusion Criteria

Child Inclusion Criteria:

1. Less than 8 days of age or previous participation in one of the BLOOM-PTN, BLOOM-LTFU, Pregnancy During the Pandemic or PROBIO studies;
2. Born at ≤ 36 weeks + 6 days gestation (36 6/7 weeks gestational age)
3. For babies recruited shortly after birth, be expected to survive more than one week;

Mother/Parent/Legal Guardian Inclusion Criteria:

1. Provide a signed and dated consent form;
2. Be able to speak and understand English;
3. Be 16 years of age or older;
4. Be willing to comply with all study procedures and be available for the duration of the study;
5. If recruited as a previous participant of the BLOOM-PTN, BLOOM-LTFU, Pregnancy During the Pandemic and/or PROBIO studies, must be willing to attend clinic visit(s) at the Alberta Children's Hospital in Calgary, Alberta at 1 and 3 years Corrected Gestational Age, or
6. If recruited within 8 days of birth, must reside within the Calgary Metropolitan Region.

Exclusion Criteria

Child Exclusion Criteria:

1. Has major congenital or chromosomal anomalies, including any congenital gastrointestinal anomalies
2. Children recruited within 8 days of birth who have a history of gastrointestinal surgery at the time of recruitment

Mother/Parent/Legal Guardian Exclusion Criteria:

1. Not the legal guardian of the child or
2. In a legal guardianship dispute.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study recruits children born premature that reside in the Calgary Metropolitan Area and their mother (where possible) parent or guardian. Children are recruited either in the first week of life or, if previously participated on at least one of the PROBIO, BLOOM PTN, Pregnancy During the Pandemic or BLOOM LTFU studies, between 3 months and 3.5 years corrected age. A control group of children born at term (≥37 weeks gestation) will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Infant outcomes at 1 and 3 years of age | 1-3.5 Years Corrected Gestational Age
  Infant outcomes as assessed by the Asthma Predictive Index, a validated methodology that helps predict asthma in young children by determining history of wheeze, atopic dermatitis, familial history and eosinophilia, and skin reactivity to common allergens via a skin prick test.

SECONDARY OUTCOMES:
Microbiome | 0-3.5 Years Corrected Gestational Age
  Microbiome establishment, fecal microbial diversity and the relative abundance of bacterial and eukaryotic taxa, as assessed by sequencing of the 16S and ITS2 gene and functional analysis via shotgun metagenomatic sequencing.
Metabolome | 0-3.5 Years Corrected Gestational Age
  Human and microbial metabolites as assessed by untargeted metabolomics, ultra-performance liquid chromatography ultrahigh-resolution Fournier transform (FT) combined with mass spectrometry.
Perinatal factors and microbiome, metabolome and immunobiome | 0-3.5 Years Corrected Gestational Age
  Influence of perinatal factors (environment, nutrition, pharmacological exposure) on the microbiome, metabolome and immunobiome; association between perinatal factors, preterm delivery, and the patterns of microbiome, metabolome and immunobiome development.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire Arrieta, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alberta BLOOM Website — http://albertabloom.ca